CLINICAL TRIAL: NCT00976391
Title: A Randomized, Open-Label, Active-Controlled, Parallel-Group, Multicenter Study to Determine the Safety and Efficacy of Albiglutide Administered in Combination With Insulin Glargine as Compared With the Combination of Insulin Glargine and Preprandial Lispro Insulin in Subjects With Type 2 Diabetes Mellitus
Brief Title: A Study to Determine the Safety and Efficacy of Albiglutide Administered in Combination With Insulin Glargine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 108486
Record Dates: First submitted 2009-09-11; First posted 2009-09-14 (Estimated); Results first posted 2014-07-16 (Estimated); Last update posted 2017-01-11 (Estimated); Status verified 2016-11

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: open-label; albiglutide; insulin glargine; preprandial insulin
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — rGLP-1 protein; Insulin Glargine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- albiglutide + insulin glargine (Active Comparator): albiglutide in combination with insulin glargine
  Interventions: Biological: albiglutide + insulin glargine
- insulin glargine + preprandial lispro insulin (Active Comparator): insulin glargine in combination with preprandial lispro insulin
  Interventions: Drug: insulin glargine + preprandial lispro insulin

INTERVENTIONS:
Biological: albiglutide + insulin glargine — albiglutide in combination with insulin glargine
  Arms: albiglutide + insulin glargine
Drug: insulin glargine + preprandial lispro insulin — insulin glargine in combination with preprandial lispro insulin
  Arms: insulin glargine + preprandial lispro insulin

SUMMARY:
This study will examine the safety and efficacy of albiglutide in combination with insulin glargine as compared with the combination of insulin glargine and preprandial lispro insulin in subjects with type 2 diabetes.

DETAILED DESCRIPTION:
This randomized, open-label, active-controlled, parallel-group, multicenter study evaluates the safety and efficacy of a weekly subcutaneously injected dose of albiglutide in combination with insulin glargine as compared with the combination of insulin glargine and preprandial lispro insulin in subjects with type 2 diabetes. Subjects with a historical diagnosis of type 2 diabetes who are inadequately controlled despite the use of insulin glargine or other intermediate- or long-acting insulins for >/= 6 months but < 5 years, with or without oral antidiabetic medications, who are unable to achieve a glycosylated hemoglobin value of < 7% will be recruited into the study. Subjects must also be willing and capable of pursuing an intensive regimen of both basal and preprandial insulin.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with type 2 diabetes, currently treated with insulin glargine or other intermediate- or long-acting insulin, with or without oral antidiabetic medications, but experiencing inadequate glycemic control and willing and capable of participating in a regimen of intensive insulin administration. A subject who has been on an intermediate- or long acting insulin for >/=6 months but <5 years, and, in spite of dosage adjustments based on home blood glucose monitoring, is unable to achieve a HbA1c of <7%.
* BMI >/= 20kg/m2 and </=45 kg/m2
* Fasting C-peptide >/=0.8 ng/mL (>/= 0.26 nmol/L)
* HbA1c between 7.0% and 10.5%, inclusive
* Use of oral or systemically injected glucocorticoids is generally not allowed within 3 months before randomization; inhaled, intra articular, and topical corticosteroids are allowed
* Hemoglobin </=11 g/dL for male subjects and >/=10 g/dL for female subjects
* Creatinine clearance >60 mL/min (calculated using the Cockcroft Gault formula)
* Thyroid stimulating hormone level is normal or clinically euthyroid as demonstrated by further thyroid tests (e.g., T4, T3, thyroid-binding globulin)
* Female subjects of childbearing potential (i.e., not surgically sterile and/or not postmenopausal) must be practicing adequate contraception. Adequate contraception must be practiced for the duration of participation in the study including the 8 week Posttreatment Follow-up Period
* Able and willing to monitor his or her own blood glucose concentrations with a home glucose monitor as per the protocol recommendations of self administration
* No major illness or debility that in the investigator's opinion prohibits the subject from actively participating in their diabetes management and completing the study
* Able and willing to provide written informed consent

Exclusion Criteria:

* History of cancer, other than squamous cell or basal cell carcinoma of the skin, that has not been in full remission for at least 3 years before Screening.
* History of treated diabetic gastroparesis
* Current ongoing symptomatic biliary disease or history of pancreatitis
* History of significant gastrointestinal surgery, including gastric bypass and banding, antrectomy, Roux en Y bypass, gastric vagotomy, small bowel resection, or surgeries thought to significantly affect upper gastrointestinal function
* Recent clinically significant cardiovascular and/or cerebrovascular disease including but not limited to the following:

  * Previous history of stroke or transient ischemic attack within 1 month before Screening.
  * Acute coronary syndrome, which includes the following:
  * Documented MI within the 2 months before Screening and during the period up until receiving the first dose of study medication
  * Any cardiac surgery including percutaneous transluminal coronary angioplasty, coronary stent placement, or coronary artery bypass graft surgery within the 2 months before Screening and during the period up until receiving the first dose of study medication
  * Unstable angina not responsive to nitroglycerin within the 2 months before Screening and during the period up until receiving the first dose of study medication
  * Unstable cardiac rhythm, however, as an example, controlled atrial fibrillation is allowed
  * Current or history of heart failure (New York Heart Association class I to IV).
  * Resting systolic pressure is >160 mm Hg and/or diastolic pressure >100 mm Hg.
  * QTc interval (Fridericia) >470 ms confirmed by a central reader at Screening
* History of stroke or other central nervous system disorder that would negatively impact the subject's ability to participate in a program of intensive insulin management (eg, physically or mentally incapable of performing home blood glucose monitoring or administering and/or adjusting insulin dosage)
* Hemoglobinopathy that may affect determination of HbA1c
* History of human immunodeficiency virus infection
* History of total bilirubin >1.5 × ULN unless the subject has a previously known history of Gilbert's syndrome and a fractionated bilirubin that shows conjugated bilirubin <35% of total bilirubin
* ALT or aspartate aminotransferase (AST) >2.5 ×ULN
* Fasting triglyceride level >850 mg/dL at Screening or Week -1 (Visit 5).
* Acute symptomatic (within 3 months before Screening) infection with hepatitis B or hepatitis C; however, subjects with past or chronic hepatitis B or hepatitis C are allowed provided the requirements for ALT, AST, and total bilirubin are met
* History of a psychiatric disorder that will affect the subject's ability to participate in the study
* History of alcohol or substance abuse within 1 year before Screening
* Positive urine drug screen at Screening, unless the subject is taking a medically approved medication for which a positive drug screen simply verifies the use of this medication
* Hypoglycemia unawareness which has impaired cognitive function and required outside assistance
* Female subject is pregnant (confirmed by laboratory testing), lactating, or <6 weeks postpartum
* Known allergy to any GLP 1 analogue, insulin, other study medications' excipients, excipients of albiglutide, or Baker's yeast
* Receipt of any investigational drug within the 30 days, or 5 half lives whichever is longer, before Screening or a history of receipt of an investigational antidiabetic drug within the 3 months before randomization, or receipt of albiglutide in previous studies
* Current use of any GLP 1 analogue
* History of type 1 diabetes mellitus, diabetic complications (e.g., active proliferative retinopathy or severe diabetic neuropathy) that in the opinion of the investigator would preclude effective participation in the study, or a history of ketoacidosis or hyperosmolar coma
* Contraindications (as per the prescribing information) for the use of either background or potential randomized study medications (e.g., insulin glargine or lispro insulin)
* History or family history of medullary carcinoma
* History or family history of multiple endocrine neoplasia type 2

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 586 (Actual)
Dates: Start 2009-09; Primary Completion 2011-10 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (180):
- United States (122):
  - GSK Investigational Site, Birmingham, Alabama
  - GSK Investigational Site, Dothan, Alabama
  - GSK Investigational Site, Gilbert, Arizona
  - GSK Investigational Site, Phoenix, Arizona
  - GSK Investigational Site, Jonesboro, Arkansas
  - GSK Investigational Site, Searcy, Arkansas
  - GSK Investigational Site, Chino, California
  - GSK Investigational Site, Commerce, California
  - GSK Investigational Site, Fresno, California
  - GSK Investigational Site, Fullerton, California
  - GSK Investigational Site, Huntington Beach, California
  - GSK Investigational Site, La Jolla, California
  - GSK Investigational Site, Long Beach, California
  - GSK Investigational Site, Los Alamitos, California
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Mission Viejo, California
  - GSK Investigational Site, Sacramento, California
  - GSK Investigational Site, San Diego, California
  - GSK Investigational Site, Satna Monica, California
  - GSK Investigational Site, Spring Valley, California
  - GSK Investigational Site, Tustin, California
  - GSK Investigational Site, Walnut Creek, California
  - GSK Investigational Site, West Hills, California
  - GSK Investigational Site, Denver, Colorado
  - GSK Investigational Site, New Britain, Connecticut
  - GSK Investigational Site, Trumbull, Connecticut
  - GSK Investigational Site, Waterbury, Connecticut
  - GSK Investigational Site, Boynton Beach, Florida
  - GSK Investigational Site, Clearwater, Florida
  - GSK Investigational Site, Cutler Bay, Florida
  - GSK Investigational Site, Hallandale, Florida
  - GSK Investigational Site, Jacksonville, Florida
  - GSK Investigational Site, Lauderdale Lakes, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Orlando, Florida
  - GSK Investigational Site, Plantation, Florida
  - GSK Investigational Site, West Palm Beach, Florida
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Blue Ridge, Georgia
  - GSK Investigational Site, Columbus, Georgia
  - GSK Investigational Site, Savannah, Georgia
  - GSK Investigational Site, Snellville, Georgia
  - GSK Investigational Site, Honolulu, Hawaii
  - GSK Investigational Site, Idaho Falls, Idaho
  - GSK Investigational Site, La Grange, Illinois
  - GSK Investigational Site, Avon, Indiana
  - GSK Investigational Site, Evansville, Indiana
  - GSK Investigational Site, Lafayette, Indiana
  - GSK Investigational Site, Council Bluffs, Iowa
  - GSK Investigational Site, Des Moines, Iowa
  - GSK Investigational Site, Iowa City, Iowa
  - GSK Investigational Site, Newton, Kansas
  - GSK Investigational Site, Topeka, Kansas
  - GSK Investigational Site, Lexington, Kentucky
  - GSK Investigational Site, Shreveport, Louisiana
  - GSK Investigational Site, Hyattsville, Maryland
  - GSK Investigational Site, Haverhill, Massachusetts
  - GSK Investigational Site, Ann Arbor, Michigan
  - GSK Investigational Site, Benzonia, Michigan
  - GSK Investigational Site, Bloomfield Hills, Michigan
  - GSK Investigational Site, Dearborn, Michigan
  - GSK Investigational Site, Kalamazoo, Michigan
  - GSK Investigational Site, Picayune, Mississippi
  - GSK Investigational Site, Chesterfield, Missouri
  - GSK Investigational Site, Jefferson City, Missouri
  - GSK Investigational Site, Kansas City, Missouri
  - GSK Investigational Site, Springfield, Missouri
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Great Falls, Montana
  - GSK Investigational Site, Omaha, Nebraska
  - GSK Investigational Site, Haddon Heights, New Jersey
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, North Massapequa, New York
  - GSK Investigational Site, Asheville, North Carolina
  - GSK Investigational Site, Burlington, North Carolina
  - GSK Investigational Site, Durham, North Carolina
  - GSK Investigational Site, Hickory, North Carolina
  - GSK Investigational Site, Morehead City, North Carolina
  - GSK Investigational Site, Tabor City, North Carolina
  - GSK Investigational Site, Akron, Ohio
  - GSK Investigational Site, Canal Fulton, Ohio
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Cleveland, Ohio
  - GSK Investigational Site, Columbus, Ohio
  - GSK Investigational Site, Dayton, Ohio
  - GSK Investigational Site, Oklahoma City, Oklahoma
  - GSK Investigational Site, Tulsa, Oklahoma
  - GSK Investigational Site, Bensalem, Pennsylvania
  - GSK Investigational Site, Carlisle, Pennsylvania
  - GSK Investigational Site, Tipton, Pennsylvania
  - GSK Investigational Site, Uniontown, Pennsylvania
  - GSK Investigational Site, Greenville, South Carolina
  - GSK Investigational Site, Murrells Inlet, South Carolina
  - GSK Investigational Site, Clarksville, Tennessee
  - GSK Investigational Site, Johnson City, Tennessee
  - GSK Investigational Site, McKenzie, Tennessee
  - GSK Investigational Site, Memphis, Tennessee
  - GSK Investigational Site, Tullahoma, Tennessee
  - GSK Investigational Site, Arlington, Texas
  - GSK Investigational Site, Bedford, Texas
  - GSK Investigational Site, Corpus Christi, Texas
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, El Paso, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, Katy, Texas
  - GSK Investigational Site, Lake Jackson, Texas
  - GSK Investigational Site, Midland, Texas
  - GSK Investigational Site, North Richland Hills, Texas
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Schertz, Texas
  - GSK Investigational Site, Sugar Land, Texas
  - GSK Investigational Site, Temple, Texas
  - GSK Investigational Site, Bountiful, Utah
  - GSK Investigational Site, Salt Lake City, Utah
  - GSK Investigational Site, South Burlington, Vermont
  - GSK Investigational Site, Burke, Virginia
  - GSK Investigational Site, Hampton, Virginia
  - GSK Investigational Site, Manassas, Virginia
  - GSK Investigational Site, Richmond, Virginia
  - GSK Investigational Site, Spokane, Washington
  - GSK Investigational Site, Tacoma, Washington
  - GSK Investigational Site, Lewisburg, West Virginia
- Brazil (3):
  - GSK Investigational Site, Porto Alegre, Rio Grande do Sul
  - GSK Investigational Site, Brasília
  - GSK Investigational Site, Mogi das Cruzes
- France (2):
  - GSK Investigational Site, Armentières
  - GSK Investigational Site, Vénissieux
- Germany (4):
  - GSK Investigational Site, Witten, North Rhine-Westphalia
  - GSK Investigational Site, Mainz, Rhineland-Palatinate
  - GSK Investigational Site, Dresden, Saxony
  - GSK Investigational Site, Berlin, State of Berlin
- GSK Investigational Site, Shatin, Hong Kong
- India (3):
  - GSK Investigational Site, Bangalore
  - GSK Investigational Site, Chennai
  - GSK Investigational Site, Manipal
- Mexico (3):
  - GSK Investigational Site, Pachuca, Hidalgo
  - GSK Investigational Site, Puebla City, Puebla
  - GSK Investigational Site, Mexico City
- Peru (5):
  - GSK Investigational Site, Ica, Ica
  - GSK Investigational Site, Lima, Lima Province
  - GSK Investigational Site, Huacho, Lima region
  - GSK Investigational Site, Piura, Piura
  - GSK Investigational Site, Trujillo
- Philippines (7):
  - GSK Investigational Site, Marikina City
  - GSK Investigational Site, Pasay
  - GSK Investigational Site, Pasig
  - GSK Investigational Site, Quezon City
  - GSK Investigational Site, San Juan City
  - GSK Investigational Site, Tagbilaran City
  - GSK Investigational Site, Taytay Rizal
- South Africa (11):
  - GSK Investigational Site, Port Elizabeth, Eastern Cape
  - GSK Investigational Site, Boksburg North, Gauteng
  - GSK Investigational Site, Johannesburg, Gauteng
  - GSK Investigational Site, Lenasia, Gauteng
  - GSK Investigational Site, Pretoria, Gauteng
  - GSK Investigational Site, Durban, KwaZulu-Natal
  - GSK Investigational Site, Bellville
  - GSK Investigational Site, Cape Town
  - GSK Investigational Site, Kempton Park
  - GSK Investigational Site, Parow
  - GSK Investigational Site, Somerset West
- South Korea (5):
  - GSK Investigational Site, Goyang-si
  - GSK Investigational Site, Koyang-shi
  - GSK Investigational Site, Seongnam-si
  - GSK Investigational Site, Seoul
  - GSK Investigational Site, Suwon, Kyonggi-do
- Spain (6):
  - GSK Investigational Site, Alzira
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Palma de Mallorca
  - GSK Investigational Site, Sabadell
  - GSK Investigational Site, Seville
- Taiwan (4):
  - GSK Investigational Site, Taichung
  - GSK Investigational Site, Tainan
  - GSK Investigational Site, Taipei
  - GSK Investigational Site, Taipei County
- United Kingdom (4):
  - GSK Investigational Site, Liverpool, Merseyside
  - GSK Investigational Site, Hull
  - GSK Investigational Site, London
  - GSK Investigational Site, Plymouth

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Rosenstock J, Fonseca VA, Gross JL, Ratner RE, Ahren B, Chow FC, Yang F, Miller D, Johnson SL, Stewart MW, Leiter LA; Harmony 6 Study Group. Advancing basal insulin replacement in type 2 diabetes inadequately controlled with insulin glargine plus oral agents: a comparison of adding albiglutide, a weekly GLP-1 receptor agonist, versus thrice-daily prandial insulin lispro. Diabetes Care. 2014 Aug;37(8):2317-25. doi: 10.2337/dc14-0001. Epub 2014 Jun 4. PMID 24898300
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Study Protocol: 108486 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 108486 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 108486 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 108486 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 108486 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 108486 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 108486 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants (par.) who met eligibility criteria and completed a 4-8 week Run-in/Stabilization Period were then randomized to a 52-week Treatment Period, followed by 8 weeks of post-treatment follow-up. A total of 920 par. were screened; 586 par. were randomized, and 566 par. received >=1 treatment dose.
Groups:
- Albiglutide 30 mg With Insulin Glargine: Participants received albiglutide 30 milligrams (mg) as a subcutaneous injection weekly (with uptitration to 50 mg weekly if needed) via a fully disposable pen injector system combined with insulin glargine (with uptitration if needed) as prescribed by their physician. Participants did not receive investigational product during the Follow-up Period.
- Preprandial Lispro Insulin With Insulin Glargine: Participants received a combination of insulin glargine (with uptitration if needed) and preprandial lispro insulin (with uptitration as appropriate) as prescribed by their physician.Participants did not receive investigational product during the Follow-up Period.
Period: Treatment Period (52 Weeks)
Arm/Group | Albiglutide 30 mg With Insulin Glargine | Preprandial Lispro Insulin With Insulin Glargine
Started | 285 | 281
Completed | 243 | 242
Not Completed | 42 | 39
Not completed — Adverse Event | 16 | 2
Not completed — Protocol Violation | 1 | 1
Not completed — Noncompliance | 4 | 4
Not completed — Lost to Follow-up | 10 | 8
Not completed — Withdrawal by Subject | 9 | 19
Not completed — Physician Decision | 1 | 1
Not completed — Termination of Study/Site by GSK | 0 | 4
Not completed — Pregnancy | 1 | 0
Period: Follow-up Period (8 Weeks)
Arm/Group | Albiglutide 30 mg With Insulin Glargine | Preprandial Lispro Insulin With Insulin Glargine
Started | 285 | 281
Completed | 256 | 247
Not Completed | 29 | 34
Not completed — Adverse Event | 3 | 1
Not completed — Noncompliance | 2 | 2
Not completed — Lost to Follow-up | 14 | 12
Not completed — Did not Entered Follow-up | 6 | 8
Not completed — Withdrawal by Subject | 4 | 7
Not completed — Termination of Study/Site by GSK | 0 | 4

BASELINE CHARACTERISTICS:
Groups:
- Albiglutide 30 mg With Insulin Glargine: Participants received albiglutide 30 mg as a subcutaneous injection weekly (with uptitration to 50 mg weekly if needed) via a fully disposable pen injector system combined with insulin glargine (with uptitration if needed) as prescribed by their physician. Participants did not receive investigational product during the Follow-up Period.
- Total: Total of all reporting groups
Arm/Group | Albiglutide 30 mg With Insulin Glargine | Preprandial Lispro Insulin With Insulin Glargine | Total
Number analyzed (Participants) | 285 | 281 | 566
Age, Continuous [Mean (Standard Deviation); unit: Years] | 54.8 (9.10) | 56.3 (8.87) | 55.6 (9.01)
Gender [Count of Participants; unit: Participants]
  Female | 153 | 145 | 298
  Male | 132 | 136 | 268
Race/Ethnicity, Customized [Number; unit: Participants] — A participant may have been counted in more than 1 category.
  Participants
    African American/African Heritage | 39 | 34 | 73
    American Indian or Alaskan Native | 29 | 20 | 49
    Asian - Central/South Asian Heritage | 17 | 17 | 34
    Asian - East Asian Heritage | 15 | 17 | 32
    Asian - South East Asian Heritage | 16 | 16 | 32
    Native Hawaiian or Other Pacific Islander | 1 | 3 | 4
    White - Arabic/North African Heritage | 2 | 3 | 5
    White - White/Caucasian/European Heritage | 174 | 171 | 345
    Other-Black | 1 | 0 | 1
    Other-Native American | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline (BL) in Glycosylated Hemoglobin (HbA1c) at Week 26
Description: HbA1c is a form of hemoglobin that is measured primarily to identify the average plasma glucose concentration over a 2- to 3-month period. The BL HbA1c value is defined as the last non-missing value before the start of treatment. Change from BL was calculated as the value at Week 26 minus the value at BL. The analysis was performed using an Analysis of Covariance (ANCOVA) model with treatment group, region, history of prior myocardial infarction (yes versus no), and age category (<65 years versus ≥65 years) as factors and Baseline HbA1c as a continuous covariate.The last observation carried forward (LOCF) method was used to impute missing post-BL HbA1c values; the last non-missing post-BL on-treatment measurement was used to impute the missing measurement. HbA1c values obtained after hyperglycemic rescue were treated as missing and were replaced with pre-rescue values.
Time Frame: Baseline and Week 26
Population: Intent-to-Treat (ITT) Population with LOCF: all randomized par. who received >=1 dose of study medication and who had a BL assessment and >=1 post-BL assessment of HbA1c. Only par. with a value at BL and at the specified visit were analyzed. Values were carried forward for par. who were rescued or discontinued from active treatment before Week 26.
Measure: Least Squares Mean (Standard Error); unit: Percentage of HbA1c in the blood
Arm/Group | Albiglutide 30 mg With Insulin Glargine | Preprandial Lispro Insulin With Insulin Glargine
Number analyzed (Participants) | 279 | 278
Percentage of HbA1c in the blood | -0.82 (0.058) | -0.66 (0.058)
Statistical Analysis 1: Comparison: Albiglutide 30 mg With Insulin Glargine vs Preprandial Lispro Insulin With Insulin Glargine; Test type: Non-Inferiority or Equivalence — P-value from a one-sided t-test to test whether the difference of least square means (albiglutide - preprandial lispro insulin) is less than or equal to the pre-specified non-inferiority margin of 0.4%; p < 0.0001, t-test, 1 sided; Mean Difference (Net) = -0.16, 95% CI 2-sided [-0.32 to 0.00]

2. Secondary Outcome: Change From Baseline in HbA1c at Weeks 36, 48 and 52
Description: HbA1c is a form of hemoglobin that is measured primarily to identify the average plasma glucose concentration over a 2- to 3-month period. Baseline is defined as the last available assessment on or prior to the first dose of study drug. Change from Baseline was calculated as the post-Baseline value minus the Baseline value. This analysis used observed HbA1c values, excluding those obtained after hyperglycemia rescue; no missing data imputation was performed.
Time Frame: Baseline and Weeks 36, 48 and 52
Population: ITT Population with observed values. Only those participants with a value at Baseline and at the specified visit were analyzed (represented by n=X, X in the category titles). Different participants may have been analyzed at different time points, so the overall number of participants analyzed reflects everyone in the ITT Population.
Measure: Mean (Standard Deviation); unit: Percentage of HbA1c in the blood
Arm/Group | Albiglutide 30 mg With Insulin Glargine | Preprandial Lispro Insulin With Insulin Glargine
Number analyzed (Participants) | 250 | 254
Percentage of HbA1c in the blood
  Week 36, n=173, 182 | -1.04 (0.990) | -0.88 (0.924)
  Week 48, n=140, 153 | -0.97 (1.070) | -0.81 (0.961)
  Week 52, n=121, 141 | -1.01 (1.024) | -0.84 (0.925)

3. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG) at Week 26
Description: The FPG test measures blood sugar levels after the participant has not eaten (fasted) for 12 to 14 hours. The Baseline FPG value is the last non-missing value before the start of treatment. The LOCF method was used to impute missing post-Baseline FPG values. FPG values obtained after hyperglycemia rescue were treated as missing and replaced with pre-rescue values. Change from Baseline was calculated as the post-Baseline value minus the Baseline value. Based on ANCOVA: change = treatment + Baseline FPG + Baseline HbA1c category + region
Time Frame: Baseline and Week 26
Population: Intent-to-Treat (ITT) Population with LOCF. Only those participants with a value at Baseline and at the specified visit were analyzed. Values were carried forward for participants who were rescued or discontinued from active treatment before Week 26.
Measure: Least Squares Mean (Standard Error); unit: Millimoles per liter (mmol/L)
Arm/Group | Albiglutide 30 mg With Insulin Glargine | Preprandial Lispro Insulin With Insulin Glargine
Number analyzed (Participants) | 282 | 279
Millimoles per liter (mmol/L) | -0.99 (0.164) | -0.71 (0.164)

4. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG) at Weeks 36, 48 and 52
Description: The FPG test measures blood sugar levels after the participant has not eaten (fasted) for 12 to 14 hours. The Baseline FPG value is the last non-missing value before the start of treatment. Change from Baseline was calculated as the post-Baseline FPG minus the Baseline FPG. This analysis used observed FPG values excluding those obtained after hyperglycemia rescue; no missing data imputation was performed.
Time Frame: Baseline and Weeks 36, 48 and 52
Population: ITT Population with observed values. Only those participants with a value at Baseline and at the specified visit were analyzed (represented by n=X, X in the category title).
Measure: Mean (Standard Deviation); unit: Millimoles per liter (mmol/L)
Arm/Group | Albiglutide 30 mg With Insulin Glargine | Preprandial Lispro Insulin With Insulin Glargine
Number analyzed (Participants) | 171 | 182
Millimoles per liter (mmol/L)
  Week 36, n=171, 182 | -1.41 (2.905) | -0.91 (3.039)
  Week 48, n=131, 151 | -1.13 (3.078) | -1.07 (2.965)
  Week 52, n=121, 139 | -1.36 (3.054) | -0.97 (3.305)

5. Secondary Outcome: Number of Participants Who Achieved HbA1c Response Level of <6.5% and <7.0% at Week 26
Description: The number of participants who acheieved the HbA1c treatment goal (i.e., HbA1c response levels of <6.5% and <7.0% at Week 26) were assessed.
Time Frame: Week 26
Population: ITT Population. Only those participants available at the indicated time point were assessed.
Measure: Number; unit: Participants
Arm/Group | Albiglutide 30 mg With Insulin Glargine | Preprandial Lispro Insulin With Insulin Glargine
Number analyzed (Participants) | 279 | 278
Participants
  HbA1c <6.5 % | 31 | 23
  HbA1c <7.0 % | 83 | 70

6. Secondary Outcome: Time to Hyperglycemia Rescue
Description: Participants who experienced persistent hyperglycemia (high blood glucose) could have qualified for hyperglycemia rescue. The conditions for hyperglycemia rescue were as follows: HbA1c >9.0% and <0.5% decrease from Baseline between >=Week 4 and <Week 8; HbA1c >9.0% and <0.5% decrease from Baseline between >=Week 8 and <Week 12; HbA1c >8.5% and >=4 weeks since uptitration between >=Week 12 and <Week 16; HbA1c >8.0% and >=4 weeks since uptitration; HbA1c >7.5% and >=4 weeks between >Week 26 and >=Week 48 since uptitration. Participants could have been rescued at any time after Week 4. Time to hyperglycemia rescue is the time between the date of first dose and the date of hyperglycemia rescue plus 1 day, or the time between the date of first dose and the date of last visit during active treatment period plus 1 day for participants not requiring rescue. This time is divided by 7 to express the result in weeks.
Time Frame: From the start of study medication until the end of the treatment (up to Week 52)
Population: ITT Population. Only those participants with a value at Baseline and at the specified visit were analyzed.
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Albiglutide 30 mg With Insulin Glargine | Preprandial Lispro Insulin With Insulin Glargine
Number analyzed (Participants) | 282 | 281
Weeks | NA [NA to NA] — There were too few events of hyperglycemia rescue (<50% of participants with events) to calculate the median and confidence interval. | NA [NA to NA] — There were too few events of hyperglycemia rescue (<50% of participants with events) to calculate the median and confidence interval.

7. Secondary Outcome: Change From Baseline in Body Weight at Week 26
Description: The Baseline value is the last non-missing value before the start of treatment. Change from Baseline was calculated as the post-Baseline weight minus the Baseline weight. The LOCF method was used to impute missing post-Baseline weight values. Weight values obtained after hyperglycemia rescue were treated as missing and replaced with prerescue values. Based on ANCOVA: change = treatment + Baseline weight + Baseline HbA1c category + prior myocardial infarction history + age category + region + current oral antidiabetic therapy.
Time Frame: Baseline and Week 26
Population: ITT Population with LOCF. Only those participants with a value at Baseline and at the specified visit were analyzed. Values were carried forward for participants who were rescued or discontinued from active treatment before Week 26.
Measure: Least Squares Mean (Standard Error); unit: Kilograms
Arm/Group | Albiglutide 30 mg With Insulin Glargine | Preprandial Lispro Insulin With Insulin Glargine
Number analyzed (Participants) | 282 | 280
Kilograms | -0.73 (0.194) | 0.81 (0.195)

8. Secondary Outcome: Change From Baseline in Body Weight at Weeks 36, 48 and 52
Description: The Baseline value is the last non-missing value before the start of treatment. Change from Baseline was calculated as the post-Baseline weight minus the Baseline weight. This analysis used observed body weight values excluding those obtained after hyperglycemia rescue; no missing data imputation was performed.
Time Frame: Baseline and Weeks 36, 48 and 52
Population: ITT Population with observed values. Only those participants who were available at the indicated time points were analyzed (represented by n=X, X in the category title).
Measure: Mean (Standard Deviation); unit: Kilograms
Arm/Group | Albiglutide 30 mg With Insulin Glargine | Preprandial Lispro Insulin With Insulin Glargine
Number analyzed (Participants) | 172 | 182
Kilograms
  Week 36, n=172, 182 | -0.42 (3.656) | 1.31 (4.005)
  Week 48, n=142, 153 | -0.60 (3.928) | 1.56 (3.846)
  Week 52, n=122, 141 | -0.70 (4.023) | 1.44 (4.053)

ADVERSE EVENTS:
Time Frame: On-treatment serious adverse events (SAEs) and non-serious adverse events (AEs), defined as those events occurring while participants were on treatment up until 56 days after the last dose (up to Week 60), are reported.
Description: SAEs and AEs were collected in members of the Safety Population, comprised of all participants randomized to treatment, who received at least one dose of the study medication.
Arm/Group | Albiglutide 30 mg With Insulin Glargine | Preprandial Lispro Insulin With Insulin Glargine
Serious Adverse Events (participants affected / at risk) | 38/285 | 29/281
Other Adverse Events (participants affected / at risk) | 188/285 | 178/281
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Albiglutide 30 mg With Insulin Glargine (N=285) | Preprandial Lispro Insulin With Insulin Glargine (N=281)
Coronary artery disease (Cardiac disorders) | 0 | 4
Acute myocardial infarction (Cardiac disorders) | 2 | 1
Angina unstable (Cardiac disorders) | 1 | 2
Atrial fibrillation (Cardiac disorders) | 2 | 0
Ventricular tachycardia (Cardiac disorders) | 1 | 1
Myocardial infarction (Cardiac disorders) | 1 | 0
Ventricular fibrillation (Cardiac disorders) | 0 | 1
Incisional hernia (Injury, poisoning and procedural complications) | 1 | 2
Road traffic accident (Injury, poisoning and procedural complications) | 2 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 0 | 1
Fibula fracture (Injury, poisoning and procedural complications) | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 1 | 0
Ligament rupture (Injury, poisoning and procedural complications) | 1 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 1
Muscle rupture (Injury, poisoning and procedural complications) | 0 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 1
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 1
Cellulitis (Infections and infestations) | 1 | 2
Abscess limb (Infections and infestations) | 0 | 1
Appendicitis (Infections and infestations) | 1 | 0
Bacterial sepsis (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 0
Gastroenteritis viral (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 1 | 0
Lobar pneumonia (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 1 | 0
Tracheobronchitis (Infections and infestations) | 1 | 0
Tuberculosis (Infections and infestations) | 1 | 0
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Ovarian germ cell teratoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Phaeochromocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pituitary tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tongue neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Chest pain (General disorders) | 1 | 2
Electrocution (General disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 1
Enterocele (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 1 | 0
Hiatus hernia (Gastrointestinal disorders) | 1 | 0
Large intestine Perforation (Gastrointestinal disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Trigger finger (Musculoskeletal and connective tissue disorders) | 1 | 0
Arteriosclerosis (Vascular disorders) | 1 | 0
Haemorrhage (Vascular disorders) | 0 | 1
Malignant hypertension (Vascular disorders) | 1 | 0
Angle closure glaucoma (Eye disorders) | 1 | 0
Diabetic retinopathy (Eye disorders) | 0 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 1
Cervical cyst (Reproductive system and breast disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0
Cholecystitis Chronic (Hepatobiliary disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Completed suicide (Psychiatric disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 0 | 1
Angioedema (Skin and subcutaneous tissue disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Albiglutide 30 mg With Insulin Glargine (N=285) | Preprandial Lispro Insulin With Insulin Glargine (N=281)
Nasopharyngitis (Infections and infestations) | 30 | 29
Urinary Tract Infection (Infections and infestations) | 29 | 27
Upper Repiratory Tract Infection (Infections and infestations) | 27 | 20
Bronchitis (Infections and infestations) | 13 | 17
Sinusitis (Infections and infestations) | 14 | 9
Influenza (Infections and infestations) | 8 | 11
Gastroenteritis (Infections and infestations) | 7 | 10
Gastroenteritis Viral (Infections and infestations) | 6 | 8
Diarrhoea (Gastrointestinal disorders) | 41 | 16
Nausea (Gastrointestinal disorders) | 37 | 6
Vomiting (Gastrointestinal disorders) | 20 | 4
Constipation (Gastrointestinal disorders) | 12 | 6
Gastritis (Gastrointestinal disorders) | 9 | 5
Gastroesophageal Reflux Disease (Gastrointestinal disorders) | 10 | 4
Dyspepsia (Gastrointestinal disorders) | 12 | 1
Abdominal Pain (Gastrointestinal disorders) | 7 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 13 | 20
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 12 | 13
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 | 12
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 13 | 4
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 8 | 7
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 6 | 5
Oedema Peripheral (General disorders) | 11 | 24
Injection Site Reaction (General disorders) | 12 | 2
Injection Site Haematoma (General disorders) | 6 | 5
Fatigue (General disorders) | 7 | 3
Diabetic Retinopathy (Eye disorders) | 18 | 23
Cataract (Eye disorders) | 11 | 9
Macular Oedema (Eye disorders) | 7 | 4
Headache (Nervous system disorders) | 21 | 12
Diabetic Neuropathy (Nervous system disorders) | 3 | 8
Hypertension (Vascular disorders) | 16 | 17
Contusion (Injury, poisoning and procedural complications) | 6 | 9
Dyslipidaemia (Metabolism and nutrition disorders) | 6 | 8
Cough (Respiratory, thoracic and mediastinal disorders) | 7 | 7
Depression (Psychiatric disorders) | 5 | 8
Ecchymosis (Skin and subcutaneous tissue disorders) | 4 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.